CLINICAL TRIAL: NCT02209922
Title: The Effects of tDCS Combined With Balance Training on Postural Control in Chronic Stroke Patients ( A Randomized Controlled Trial)
Brief Title: The Effects of tDCS Combined With Balance Training on Postural Control in Chronic Stroke Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fariba Yadolahi, Fariba Yadolahi-MD-MPH-PhD Candidate in physical therapy, Shahid Beheshti University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tDCS and postural control; 15840 (Other: Shahid Beheshti University of Medical Sciences-IRAN)
Record Dates: First submitted 2014-07-30; First posted 2014-08-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Ischemic Stroke
Keywords: tDCS, stroke, postural control
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial direct current stimulation (Active Comparator): ARM1: Transcranial direct current stimulation (tDCS) intervention and simultaneous balance training.
  Participants underwent tDCS(2mA) brain stimulation (20 minutes) and simultaneous balance training(20 minutes) for 5 consecutive days,for 1 week.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- ARM 2 (Sham Comparator): ARM2: Sham tDCS and simultaneous balance training(20 minutes) for 5 consecutive days,for 1 week.
  Interventions: Device: Sham

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — Participants underwent tDCS(2mA) brain stimulation (20 minutes) and simultaneous balance training(20 minutes) for 5 consecutive days,for 1 week.
  Arms: Transcranial direct current stimulation
Device: Sham — During sham stimulation, the current ramped up for 30 seconds, ramped back down for 30 seconds, and then remained off for the duration of the stimulation then and simultaneous balance training(20 minutes) for 5 consecutive days,for 1 week.
  Arms: ARM 2

SUMMARY:
Purpose:

The incidence of stroke in low-to-middle income countries is increasing .Balance impairment and falling negatively impact function of stroke patients. Mobility is based on successful postural control and about 30% of individuals with stroke are unable to ambulate without assistance.Transcranial direct current stimulation (tDCS) is a new promising tool for motor recovery in neurological disease.This can be addressed through a tDCS intervention.

Objective:The objectives of this study is to examine the efficacy of anodal tDCS combined with Biodex balance training on postural control in chronic stroke patients using laboratory and clinical assessments. The following essential treatment components; a) active tDCS stimulation paired with Biodex balance training, b)sham tDCS paired with Biodex balance training program.

To identify combinations effects of tDCS stimulation plus balance training . Hypothesis: Anodal tDCS targeting leg motor area (CZ) for 5-days plus Biodex balance training, will significantly improve stroke clients' balance and functional mobility.

Double blinded sham -controlled randomized tDCS stimulation Arms Assigned Interventions

Experimental: Arm 1

tDCS brain stimulation and simultaneous balance training

Participants underwent Active tDCS brain stimulation (20 minutes) and simultaneous balance training(20 minutes) for 5 consecutive days.

No Intervention: Arm 2 Sham tDCS brain stimulation (20 minutes) and simultaneous balance training

DETAILED DESCRIPTION:
Participants underwent tDCS(2mA) brain stimulation (20 minutes) and simultaneous balance training(20 minutes) for 5 consecutive days, All outcome measures will be measured in 4 time points: pre-test, post-test after 10 sessions of intervention, and after 1 week and 1 months post intervention as follow ups.

ELIGIBILITY:
Inclusion Criteria:

age ≥18 years; first-ever ischemic stroke; chronic phase of recovery (>6 months); ability to walk 6- meter supported or unsupported; ability to stand at least unsupported for 40-seconds with eyes closed; only ischemic stroke involving middle cerebral artery (MCA) territory confirmed by CT or MRI.

Exclusion Criteria:

Use of any neuro- or psycho-active medications that alters balance; any other neurological conditions or sensory disorders affecting postural control; such as brain tumor, or substance abuse; orthopedic diseases; ongoing/recent (within 3 months) balance rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-12; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Postural control | After 5 days
  Functional dynamic balance

SECONDARY OUTCOMES:
Static Balance | After 5 days
  linear analysis
Change of Static Balance | 1 week
  linear analysis
Change of Static Balance | 1 month
  linear analysis

OTHER OUTCOMES:
Postural sway flactuation | After 5 days
  nonlinear (Approximate entropy) analysis
Postural sway flactuation | 1 week
  nonlinear (Approximate entropy) analysis
Postural sway flactuation | 1 month
  nonlinear (Approximate entropy) analysis
Change of Postural control | 1 week
  Functional dynamic balance
Change of Postural control | 1 month
  Functional dynamic balance

CONTACTS AND LOCATIONS:
Overall Officials: Fariba Yadolahi, MD-MPH-PhD, Principal Investigator — Department of Physical therapy-School of Rehabilitation-Shahid Beheshti University of Medical sciences
Locations (1):
- Shahid Beheshti Univesity of Medical sciences, Tehran, Iran

REFERENCES:
- [Derived] Elsner B, Kugler J, Pohl M, Mehrholz J. Transcranial direct current stimulation (tDCS) for improving activities of daily living, and physical and cognitive functioning, in people after stroke. Cochrane Database Syst Rev. 2020 Nov 11;11(11):CD009645. doi: 10.1002/14651858.CD009645.pub4. PMID 33175411